CLINICAL TRIAL: NCT01326221
Title: Extracellular and Intracellular TFV/FTC Residues After a Single Dose in HIV-Negative Men and Women: Implications for Pre-exposure HIV Prophylaxis Dosing of Truvada®
Brief Title: Single Dose Truvada in HIV-negative Men and Women
Acronym: TAIL
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Angela Kashuba, PharmD, Professor, University of North Carolina, Chapel Hill
Other Study IDs: 08-0410
Record Dates: First submitted 2009-03-02; First posted 2011-03-30 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Pharmacokinetic Study in Healthy Volunteers
Keywords: Truvada; tenofovir; emtricitabine; Pharmacokinetics; Healthy Volunteers
MeSH Terms: interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Single dose of Truvada
  Interventions: Drug: tenofovir + emtricitabine

INTERVENTIONS:
Drug: tenofovir + emtricitabine — tenofovir 300mg + emtricitabine 200mg x one dose
  Other Names: Truvada

SUMMARY:
This open-label, non-blinded, pharmacokinetic (PK) study will assess both tenofovir and emtricitabine (components of Truvada) concentrations within genital tract of male and females after a single dose of Truvada®. Concentrations of the active drug will be measured in blood (women and men), cervicovaginal aspirates and vaginal tissue (women only), seminal fluid and rectal tissue (men only). Samples will be obtained at 24 hours (1 day), 48 hours (2 days), 5 days, 7 days, 10 days, and 14 days post-dose. Each subject will undergo 2 biopsy days, at least 72 hours apart. Additionally, tissue samples will be evaluated ex-vivo for HIV infectivity.

DETAILED DESCRIPTION:
An estimated 80% of HIV infections worldwide are acquired through sexual transmission.1 Viable methods of preventing the sexual transmission of HIV are urgently needed, especially in resource-poor countries. As these countries now have increased access to generic antiretroviral medications, oral administration of antiretroviral drugs as pre-exposure prophylaxis may serve as a feasible, minimally invasive mechanism of preventing the sexual transmission of HIV globally.

Antiretroviral prophylaxis with the combination of tenofovir and emtricitabine has recently been investigated by the U.S. Centers for Disease Control and Prevention in a series of studies with rhesus macaques. Researchers developed a rectal inoculation model using concentrations of Simian HIV (SIV) that were representative of HIV exposure in humans. With this model, researchers demonstrated that standard doses of tenofovir disoproxil fumarate delayed, or partially protected, animals from the acquisition of Simian HIV during a 14-week time period. In this same model, high dose tenofovir was fully protective from infection.2 However, it is unknown how concentrations in the macaque mucosal surfaces compare to that in humans. Notwithstanding, a number of clinical studies are currently investigating daily dosing of tenofovir or tenofovir with emtricitabine for pre-exposure prophylaxis.3

Since daily dosing of antiretrovirals for pre-exposure prophylaxis is not sustainable long-term, other coitally-dependent (episodic) dosing strategies are needed. However, the extent to which these drugs concentrate in tissues, and the duration of intracellular phosphate exposure after single doses, is currently unknown. This information is required to inform the potential of success with these dosing strategies.

At steady-state concentrations, the mean blood plasma half-life (t½) of tenofovir and emtricitabine are 15.9 hours and 10.7 hours, respectively. 4 However, the intracellular t½ of tenofovir diphosphate and emtricitabine triphosphate are >60 hours and 39 hours, respectively.5 The long intracellular t½ of the active forms of these drugs might hold advantages for episodic dosing. However, the long t½ might also hold disadvantages in terms of the development of viral resistance mutations. This phenomenon (the development of resistance after a single dose of a long t½ drug), has been previously seen with nevirapine given during delivery to HIV-infected women to prevent mother to child transmission of HIV.6 However, these women were chronically infected, rather than newly infected, as would be the case with populations exposed to prevention strategies.

The proposed study aims to augment the information gathered in previous studies by examining intracellular and extracellular tenofovir and emtricitabine drug concentrations in various human compartments after a single dose, and to describe the potential for HIV infectivity in selected tissue samples obtained from these compartments.

ELIGIBILITY:
Inclusion Criteria:

* Must be above 18 years of age and less than 50 years of age
* Able and willing to provide written informed consent to take part in the study
* Able and willing to provide adequate information for locator purposes
* Must be in good general health by volunteer history without any clinically significant systemic disease, full physical examination including blood pressure and pulse rate measurement and clinical laboratory tests
* HIV-1 status antibody negative as documented at screening
* Able to comply with all study procedures throughout the duration of study participation
* Able to comply with Lifestyle Guidelines throughout the duration of study participation

(Males Only)

* Willing to abstain from any sexual activity including intercourse, masturbation, oral contact with the rectum, and insertion of anything per rectum for the entire duration of the study period.
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight > 50 kg (110 lbs).

(Females Only)

* Must be pre-menopausal
* Must have an intact uterus and cervix
* Must have a negative serum pregnancy test at screening
* Must have negative urine pregnancy tests at day 7 and day 14
* Must have regular menstrual cycles (minimum of 26 and maximum of 35 days)
* Must be at least 2 months since last pregnancy outcome and have had at least two spontaneous menses
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight > 50 kg (110 lbs).
* Must abstain from use of intravaginal products including tampons, spermicides, lubricants, vaginal hygiene products, diaphragms, and cervical caps, for 72 hours prior to the baseline study visit and through 21 days after the baseline study visit.
* Must abstain from any sexual activity including intercourse, oral contact with the female genitalia, masturbation, and penetration of the vagina by fingers, tampons, sex toys, or any other objects for 72 hours prior to the baseline study visit (Day 0) and through 19 days after the baseline study visit.

Exclusion Criteria:

* HIV positive at screening
* A positive result for Hepatitis B surface antigen (HbsAg) or Hepatitis B core antibody (HbcAb) screening tests or anti-hepatitis C virus serology (as determined by multi-antigen EIA)
* Active infection at the time of entry
* Active sexually transmitted disease(s)
* History of abnormal bleeding or bruising
* History of kidney disease
* History of alcoholism or drug abuse
* History of significant gastrointestinal bleeding
* History of severe or recent cardiac or pulmonary event
* Use of prescription or non-prescription drugs, vitamins, and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the baseline study visit day.
* Use of herbal supplements within 14 days of the baseline study visit day.
* Treatment with an investigational drug within 4 months preceding the baseline study visit day.
* Unwillingness to refrain from chronic use of aspirin and NSAIDS
* > Grade 2 laboratory abnormality
* Any other clinical condition or therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
* Unwilling or unable to comply with the lifestyle guidelines for the entire duration of study participation. The lifestyle guidelines are outlined in Appendix A.
* Allergy to local anesthetics (lidocaine) or silver nitrate or iron-containing substances

(Males Only)

* Active rectal infection at screen
* History of inflammatory bowel disease
* History or symptoms of gastrointestinal disease

(Females Only)

* Currently pregnant or at risk for pregnancy (may be using Paragard® IUD, effective barrier method, female sterilization or abstinence, or be sexually active with a vasectomized partner)
* Currently breastfeeding
* Positive test for Neisseria gonorrhoea, Chlamydia trachomatis, Trichomonas vaginalis or syphilis at screen.
* Use of any hormonal contraceptives within 30 days of enrollment.
* Use of Depo-Provera within 120 days of enrollment.
* Current vaginal or urinary tract infection

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twelve adult (18 years or older) healthy volunteers will be recruited to participate in the study. A total of 6 men and 6 women will be enrolled. Subjects of all races and ethnicities may participate, provided they meet study inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
TFV, TFV-DP, FTC, FTC-TP in blood, CVF, cervical and vaginal and rectal tissue over 14 days | 14 days
  The study aims to examine intra- and extracellular tenofovir and emtricitabine concentrations in various human compartments after a single dose, and to look at the potential for HIV infectivity in tissue samples from these compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina; Kristine B Patterson, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States